CLINICAL TRIAL: NCT05446155
Title: BioMEL - a Translational Study About Aetiology, Diagnosis, Prognosis, Treatment, Biology and Biomarkers in Clinically Atypical Nevi and Melanoma.
Brief Title: BioMEL- Diagnostic and Prognostic Factors in Melanoma.
Acronym: BioMEL
Status: Recruiting | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-101
Record Dates: First submitted 2022-07-01; First posted 2022-07-06 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Melanoma; Melanoma in Situ; Dysplastic Nevi; Mole (Dermatology); Image; Mutation
Keywords: Biobank; Melanoma; nevus; mole; dermoscopy; dermatoscopy; skin cancer; Sequence analysis, DNA; Sequence analysis, RNA; Whole genome sequencing
MeSH Terms: conditions — Melanoma; Dysplastic Nevus Syndrome; Nevus; Skin Neoplasms | interventions — Diagnostic Imaging; Genome; Dermoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples, tumour tissue samples (1 mm punch biopsy) from the primary tumour and normal, adjacent skin (2 mm punch biopsy). Tissue biopsies from melanoma metastases (excisional/punch biopsy)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with a suspected primary melanoma or equivocal pigmented skin tumour: Patients, 18 years or older, in dermatological outpatient routine care in Helsingborg, Lund or Malmö Hospitals. Patients are planned for surgical excision for an equivocal pigmented skin lesion that could be a primary melanoma or a differential diagnosis of melanoma. Imaging of tumours will be applied before surgery. Blood samples are taken before surgery. Tumour/normal skin biopsies will be taken and snap-frozen (-80°C) immediately after surgery. A baseline questionnaire about skin cancer risk factors, co-morbidities, phenotypic factors, diets, smoking, alcohol and quality of life will be given to the patient before surgery.
  Interventions: Diagnostic Test: Imaging
- Patients with secondary melanoma (metastatic disease): Patients, 18 years or older, in surgical or oncological routine care in Helsingborg, Lund, Malmö or Kristianstad Hospitals. Patients are planned for surgical excision or cytological diagnostics (needle aspiration) of metastatic melanoma. Imaging of tumours will be applied before surgery. Blood samples are taken before surgery. Tumour biopsies will be taken and snap-frozen (-80°C) immediately after surgery. A baseline questionnaire about skin cancer risk factors, co-morbidities, phenotypic factors, diets, smoking, alcohol and quality of life will be given to the patient before surgery.
  Interventions: Diagnostic Test: Imaging

INTERVENTIONS:
Diagnostic Test: Imaging — Diagnostic and prognostic imaging, omics and machine learning methods will be applied
  Other Names: transcriptomics; genomics; metabolomics; histopathological examination; deep and spatial sequencing; dermoscopy; machine learning methods

SUMMARY:
The investigators' hypothesis is that cutaneous melanoma, melanoma in situ, dysplastic nevi and benign nevi all differ in not only clinical characteristics but also molecular and genotypic characteristics.

Patients with suspected primary cutaneous melanoma or a differential diagnosis, or secondary melanoma can be asked to participate in the first part of the project and patients with suspected or confirmed secondary (spread) melanoma can be included in the second part of the study. Participants included in the study answer a validated questionnaire regarding epidemiological and phenotypic factors to map medical history, prior UV exposure, family history of melanoma and/or other cancer types, skin type, smoking habits, alcohol use and quality of life.

Blood samples (whole blood) are collected before primary local excision and before secondary surgical procedures as well as during follow up of patients with secondary disease and oncologic treatment. During local excision of the primary pigmented skin lesion, full-thickness skin punch biopsies are taken by trained dermatologists. The biopsies, in the lesion and next to the lesion in the normal skin of the suspected melanoma, are taken, snap frozen and stored deep frozen. The primary lesions are documented by accurate imaging methods prior to excision.

Tissue samples from suspected or confirmed secondary melanomas are collected mainly through surgical and core needle biopsies before, during and after treatment and in case of disease progress or treatment failure. Tissue samples are snap-frozen and stored in the same way as samples from primary melanomas.

Comprehensive questionnaire based, imaging-based information, as well as histologic information provided from the pathologist report is included and stored in a secure database.

All the information in the database, along with information from molecular analysis of tissue and/or blood samples will then be used to find objective, molecular and clinical differences in melanoma, melanoma in situ, dysplastic and benign nevi along with potential information of biological aggressivity of both primary and secondary melanoma in order to find more objective diagnostic markers.

DETAILED DESCRIPTION:
See above.

ELIGIBILITY:
Inclusion Criteria:

* Primary part of the project: Patients in dermatological outpatient routine care in Helsingborg, Lund or Malmö Hospitals. Patients are planned for surgical excision for an equivocal pigmented skin lesion that could be a primary melanoma or a differential diagnosis of melanoma
* Secondary part of the project: . Patient, in surgical or oncological routine care in Helsingborg, Lund, Malmö or Kristianstad Hospitals. Patients are planned for surgical excision or cytological diagnostics (needle aspiration) of metastatic melanoma.
* All subjects have to be able to provide written informed consent.

Exclusion Criteria:

* Patients with lesions, primary or secondary, that are so small that a punch biopsy for the study would risk affecting the histopathological diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants, clinical patients, recruited in the Southern Swedish health care region, Region Skane. Patients are recruited in the daily clinical practices in the departments of Dermatology, Surgery (including, ENT, Neuro, General surgery, Gynecology) and Oncology.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2013-11-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Genomic and transcriptomic differences between cutaneous melanoma, melanoma in situ, dysplastic nevi and benign nevi. | Cross sectional (subjects included november 2013- december 2026.
  Genomic and transcriptomic differences as analysed from DNA and RNA collected from tumour tissue biopsies from cutaneous melanoma, melanoma in situ, dysplastic nevi and benign nevi.
Interindividual genomic and transcriptomic differences in metastatic melanoma | Cross sectional (subjects included november 2013- december 2026.
  Genomic and transcriptomic differences as analysed from DNA and RNA collected from tumour tissue biopsies from metastatic melanoma.

CONTACTS AND LOCATIONS:
Overall Officials: Kari Nielsen, Ass. Prof., Principal Investigator — Lund University Cancer Centre
Locations (4):
- Sweden (4):
  - Helsingborg Hospital, Helsingborg, Skåne County
  - Kristianstad Hospital, Kristianstad, Skåne County
  - Lund University Hospital, Lund, Skåne County
  - Skåne University Hospital Malmö, Malmo, Skåne County

IPD SHARING:
Plan to Share IPD: No
For now, only researchers involved in the project can access the data, but this can change after completion of the data gathering.

REFERENCES:
- [Derived] Helkkula T, Christensen G, Ingvar C, Isaksson K, Harbst K, Persson B, Ingvar A, Hafstrom A, Carneiro A, Gaspar V, Jonsson G, Nielsen K. BioMEL: a translational research biobank of melanocytic lesions and melanoma. BMJ Open. 2024 Feb 2;14(2):e069694. doi: 10.1136/bmjopen-2022-069694. PMID 38309755
- See also: BioMEL home page — https://biomel.org/english